CLINICAL TRIAL: NCT06245837
Title: Multicenter, Non-interventional, Observational Study of Treatment and Biomarker Testing Patterns, Treatment Outcomes in Advanced/Metastatic NSCLC With and Without Actionable Genomic Alterations in Routine Clinical Practice in Russia
Brief Title: Treatment and Biomarker Testing Patterns,Treatment Outcomes in a/m NSCLC With and Without Actionable Genomic Alterations
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00204
Record Dates: First submitted 2024-01-18; First posted 2024-02-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Planned study population consists of approximately 1500 adult patients with a/m NSCLC in Russia, in about 20 oncological centers (in each center it is expected to recruit about 75 patients) in different regions of Russia in order to provide representative study sample

ELIGIBILITY:
Inclusion Criteria:

1. Morphologically confirmed NSCLC with or without actionable genomic alterations (AGA, i.e. EGFR, ALK, ROS1, NTRK, BRAF, MET exon 14 skipping, RET, ERBB2 (HER2), or KRAS)
2. Age ≥18 years at the time of NSCLC diagnosis;
3. Locally advanced or metastatic disease defined as incident stage IIIB/IIIC/IV NSCLC or stage I-IIIA then progressed to stage IIIB-IV disease and not eligible for curative-intent treatment (the date of progression is included in the database);
4. Available data on at least one line of systemic therapy for advanced/metastatic disease within the period since January 2022 until January 2025;
5. Patients may be alive or deceased at the time of medical record abstraction

Exclusion Criteria:

1. Patients participated or participating in clinical trials or any early access program within period since the index date until the end of study period;
2. Diagnosis of another cancer (except for melanoma/skin cancer) at or within 5 years prior to NSCLC diagnosis or any ongoing systemic anti-cancer therapy regimen at the time of NSCLC diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of patients with a/m NSCLC with available data on at least one line of systemic therapy for advanced/metastatic disease within the period since January 2022 until January 2025.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess treatment patterns in advanced/metastatic NSCLC in Russia and its change over time. | 12 months
  Treatment patterns after prescription of sequential/concurrent immunotherapy +/- platinum-based chemotherapy for non-AGA / AGA patients;

SECONDARY OUTCOMES:
To analyze demographic characteristics of patients with NSCLC treated in Russian oncology centers | 12 months
  Mean age at the time of a/m NSCLC diagnosis;
To assess biomarker testing patterns in advanced/metastatic NSCLC | 12 months
  PD-L1 expression status
To analyze clinical characteristics of patients with NSCLC treated in Russian oncology centers | 12 months
  Proportion of patients with de novo and recurrent advanced/metastatic disease

OTHER OUTCOMES:
To describe patient tolerability issues associated with chemotherapy in second and subsequent lines of therapy | 12 months
  Percentage of adverse events associated with chemotherapy in second and subsequent lines of therapy

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Irkutsk
  - Research Site, Kemerovo
  - Research Site, Kostroma
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Novokuznetsk
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Perm
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Vladivostok
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home